CLINICAL TRIAL: NCT06485791
Title: Evaluation of the Variation of the Intestinal Microbiota and the Integrity of the Intestinal Barrier in Patients With M.D.R. Germ-induced Pneumonia Undergoing Enteral Nutrition
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Russo Francesco, MD (Unknown); Rossella Donghia, Biologist (Unknown); Maria Notarnicola, Clinical Pathology Director (Unknown); Pasqua Letizia Pesole, Biologist (Unknown); Sergio Coletta, Laboratory Technician (Unknown); Anna Ancora, Laboratory Technician (Unknown); Francesco Gabriele, Intensive Care Unit Director (Unknown)
Responsible Party: Principal Investigator, Dr. Nicola Cappellano - MD, Principal Investigator, MD, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: MDR&Microbiota
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Multi Drug Resistant; Dysphagia
Keywords: Antibiotic resistance; Enteral nutrition
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Feces, serum, urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate the effects of enteral nutrition in subjects with MDR on the intestinal microbiota

DETAILED DESCRIPTION:
The M.D.R. it is defined as multiple resistance to antibiotics and its prevalence in intensive care units (ICU) is continuously increasing throughout the world, with great variability between continents, but also between the microorganisms themselves involved. It is estimated that global mortality attributable to antibiotic resistance is approximately 1.3 million deaths/year.

The study in question is a prospective observational study in which the effect of enteral nutrition in patients suffering from MDR on the intestinal microbiota will be evaluated. This study will enroll patients who will be hospitalized at the Resuscitation Center in the U.O.C. of Anesthesia and Resuscitation and Intensive Care of our institution, after having been admitted to other hospitals following a traumatic event which required mechanical ventilation.

Following tracheostomy, patients developed an infection detected by tracheobronchial aspirate The infection was subsequently treated with high doses of various antibiotics which led to the onset of pneumonia caused by M.D.R. germs.

Once the overall clinical picture has stabilized, i.e. the specialist needs have ceased, patients come to the U.O.C. of Anesthesia and Intensive Care Unit with a clinical picture compromised by the use of antibiotics, which caused a modification of the intestinal bacterial flora and microbiota. In fact, these patients present soft or liquid stools, as well as persistent diarrhea. Therefore they are hospitalized to proceed with nutritional rehabilitation using Enteral Nutrition, as they are very often dysphagic and therefore unable to feed themselves independently, and consequently "wash out" of antibiotics from the moment of transfer.

As per normal clinical practice, enteral nutrition is started for these patients to avoid the risk of malnutrition. For the purpose of standardizing the study, three different commercial formulations of enteral nutrition are used depending on the presence or absence of concomitant pathologies:

* Jevity Plus from the Abbot company for patients who do not have prevalent pathologies;
* Oxepa from the Abbot company for patients presenting with acute pneumonia;
* Novasource Gi Balance from the Nestlé company for diabetic patients in whom glycemic control is necessary due to diabetes mellitus.

Treatment with enteral nutrition lasts 10 days, at the end of which patients are discharged or, alternatively, leave the study.

For this study, the investigators will collect stool, urine, and serum samples for analysis of the fecal microbiota and metabolome and assessment of intestinal barrier integrity.

After signing the informed consent by the patient or by a close relative/legal representative (in the hypothesis that the patient is incapable of signing the consent), the investigator will proceed with the collection of the samples.

The samples will be collected at V0 upon admission, i.e. before starting artificial enteral nutrition, and at V1, i.e. after 10 days of enteral nutritional administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Intensive Care Unit suffering from lung infections caused by M.D.R. germs.

Exclusion Criteria:

* Patients hospitalized with other pathologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients who will be hospitalized in the U.O.C. of Anesthesia and Intensive Care of our institution, after having been admitted to other hospitals following a traumatic event which required mechanical ventilation.
  Following tracheostomy, patients developed an infection. The infection was subsequently treated with high doses of various antibiotics which led to the onset of pneumonia caused by M.D.R. germs.
  Once the overall clinical picture has stabilized, i.e. the specialist needs have ceased, patients come to the U.O.C. of Anesthesia and Intensive Care Unit with a clinical picture compromised by the use of antibiotics, which caused a modification of the intestinal bacterial flora and microbiota. Therefore they are hospitalized to proceed with nutritional rehabilitation using Enteral Nutrition, as they are very often dysphagic and therefore unable to feed themselves independently, and consequently "wash out" of antibiotics from the moment of transfer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Composition of the microbiota | at Baseline and after 10 days
  Improvement in the composition of the intestinal microbiota. Characterization of the microbiome will be carried out using a DNA metabarcoding and shotgun metatranscriptomics approach. DNA metabarcoding analysis will be conducted using the V5-V6 hypervariable regions of 16S rRNA for bacteria (MiSeq-Illumina platform). Samples found significant at DNA metabarcoding analysis will be subjected to metatracriptomic analysis (NextSeq 500 platform-Illumina). Metagenomic and metatracriptomic data will be analyzed using bioinformatics pipelines.

SECONDARY OUTCOMES:
Evaluation of the integrity of the intestinal barrier | at Baseline and after 10 days
  Improved intestinal barrier function and integrity, assessed by measuring fecal zonulin and indole and skatole by elisa technique

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Cappellano, MD, Principal Investigator — Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis

REFERENCES:
- [Background] Han Y, Zhang J, Zhang HZ, Zhang XY, Wang YM. Multidrug-resistant organisms in intensive care units and logistic analysis of risk factors. World J Clin Cases. 2022 Feb 26;10(6):1795-1805. doi: 10.12998/wjcc.v10.i6.1795. PMID 35317164
- [Background] Kent AG, Vill AC, Shi Q, Satlin MJ, Brito IL. Widespread transfer of mobile antibiotic resistance genes within individual gut microbiomes revealed through bacterial Hi-C. Nat Commun. 2020 Sep 1;11(1):4379. doi: 10.1038/s41467-020-18164-7. PMID 32873785
- [Background] Dubourg G, Lagier JC, Robert C, Armougom F, Hugon P, Metidji S, Dione N, Dangui NP, Pfleiderer A, Abrahao J, Musso D, Papazian L, Brouqui P, Bibi F, Yasir M, Vialettes B, Raoult D. Culturomics and pyrosequencing evidence of the reduction in gut microbiota diversity in patients with broad-spectrum antibiotics. Int J Antimicrob Agents. 2014 Aug;44(2):117-24. doi: 10.1016/j.ijantimicag.2014.04.020. Epub 2014 Jun 14. PMID 25063078